CLINICAL TRIAL: NCT07358468
Title: Effects Of Endometrial Preparation Protocols On Peristalsis And Pregnancy Rates In Frozen Embryo Transfer: A Prospective Cohort Study
Brief Title: Impact Of FET Preparation Protocol On Endometrial Peristalsis: A Prospective Cohort Study
Acronym: EPFE
Status: Not yet recruiting | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Collaborators: My Duc Phu Nhuan Hospital HCMC, Vietnam (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18/25/DD-BVMD
Record Dates: First submitted 2025-12-26; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Infertility; Endometrial Peristalsis; Uterine Contraction; Endometrial Waves; Frozen Embryo Transfer (FET); Uterine Peristalsis
Keywords: endometrial peristalsis; uterine contractions; endometrial waves; frozen embryo transfer; natural cycles; artificial cycles
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exogenous steroid protocol: The endometrium was prepared with the use of oral estradiol valerate (Progynova®; Delpharm Lille SAS, France, or Valiera®, Laboratorios Recalcine) at a dose of 6 mg per day, starting on the second, third, or fourth day of the menstrual cycle. Endometrial thickness was monitored from day 10 onward, and vaginal progesterone (Cyclogest, LD Collins, UK) at a dose of 800 mg per day and dydrogesterone (Duphaston, Abbott Biologicals B.V, US) at a dose of 20 mg per day were started when the endometrial thickness reached 8 mm or more. Embryo transfer was performed at 4 days for cleavage embryos transfer or 6 days for blastocyst embryo transfer after starting progesterone. All embryos were warmed on the day of transfer. Vaginal progesterone administration will be maintained until the day of the pregnancy test. In the event of a positive test result, luteal phase support will be extended until 10 weeks of gestation.
  Interventions: Other: Endometrial peristalsis and hormone measurements
- Natural protocol (True natural cycle or modified natural cycle): Daily ultrasound and serum estradiol and LH level evaluation will be performed when the mean diameter of the dominant follicle of ≥14 mm. On natural cycle, LH surge initiation is defined as a concentration of 180% above the latest serum value available in that patient with a continued rise thereafter to a level of 20 IU/l or more detected by the ECLIA method (Roche Cobas® E 801, Roche Diagnostics, Germany). On modified natural cycle, when the mean diameter of the dominant follicle is ≥16 mm, human chorionic gonadotropin (hCG, Ovitrelle® 250 µg; Merck, USA) will be injected to trigger ovulation. Vaginal progesterone (Cyclogest, LD Collins, UK) at a dose of 800 mg per day was started 2 days after the LH surge/ hCG injection. Embryo transfer will be scheduled by the time of the initiation of LH and embryo stages. Vaginal progesterone administration will be maintained until the day of the pregnancy test. In the event of a positive test result, luteal phase
  Interventions: Other: Endometrial peristalsis and hormone measurements

INTERVENTIONS:
Other: Endometrial peristalsis and hormone measurements — Time point for measurement
  Endometrial peristalsis will be assessed at three specific time points:
  * On the second day to the fourth day of the menstrual cycle in the FET cycles.
  * The day of progesterone initiation or LH surge/hCG trigger, (before progesterone exposure)
  * On the day of embryo transfer, immediately prior to the procedure
  Hormone measurements
  Serum levels of estradiol (E2) and progesterone (P4) will be assessed three times, on the same days as the endometrial peristalsis measurements, using electrochemiluminescence immunoassays. (Elecsys® Estradiol III and Elecsys® Progesterone III, Cobas® e 411, Roche Diagnostics, Germany):
  * On the second day to the fourth day of the menstrual cycle in the FET cycles
  * The day of progesterone initiation or LH surge/hCG trigger
  * On the transfer day prior to the procedure.

SUMMARY:
The uterus is a dynamic muscular organ that undergoes rhythmic, wave-like contractions known as endometrial peristalsis or endometrial waves. This muscular activity, which is an essential component of natural fertility, presents a nuanced and sometimes contradictory role in the context of assisted reproductive treatments. Endometrial peristalsis refers to the frequency, amplitude, and pattern of myometrial contractions occurring in different reproductive phases. These peristalsis play vital roles in sperm transport, embryo migration, and implantation. Clinical and imaging studies suggest that abnormal patterns or excessive contractility at the time of embryo transfer may disrupt endometrial-embryo synchrony, impair implantation, and increase miscarriage risk. However, most evidence on endometrial peristalsis pertains to fresh embryo transfer cycles, natural conceptions, or pathological contexts, such as adenomyosis or fibroids, with limited insights regarding its effects on different endometrial preparation protocols in frozen embryo transfer (FET). Understanding the dynamics of endometrial peristalsis in this context is clinically important, as inappropriate contractile activity could physically expel the embryo or create a non-receptive environment, ultimately reducing the chances of live birth. Despite its theoretical significance, there is a paucity of robust, prospective data correlating endometrial peristalsis patterns measured around the time of FET with different endometrial preparation protocols with subsequent pregnancy outcomes.

DETAILED DESCRIPTION:
The uterus is a dynamic muscular organ that undergoes rhythmic, wave-like contractions known as endometrial peristalsis or endometrial waves. This muscular activity, which is an essential component of natural fertility, presents a nuanced and sometimes contradictory role in the context of assisted reproductive treatments. Endometrial peristalsis refers to the frequency, amplitude, and pattern of myometrial contractions occurring in different reproductive phases. These peristalsis play vital roles in sperm transport, embryo migration, and implantation.

Clinical and imaging studies suggest that abnormal patterns or excessive contractility at the time of embryo transfer may disrupt endometrial-embryo synchrony, impair implantation, and increase miscarriage risk. However, most evidence on uterine contractility pertains to fresh embryo transfer cycles, natural conceptions, or pathological contexts, such as adenomyosis or fibroids, with limited insights regarding its effects on different FET protocols. Several studies have demonstrated an inverse relationship between endometrial peristalsis and IVF success. Masroor et al. found that patients with lower endometrial peristaltic wave frequency (<4 waves/min) before embryo transfer had significantly higher chances of clinical pregnancy and live birth compared to those with more frequent peristalsis. Similarly, Chung et al. reported that increased endometrial peristalsis frequency immediately after embryo transfer was linked to reduced live birth rates, suggesting that excessive motility may physically expel the embryo or disturb its implantation. In the prospective cohort study of 292 infertile women, Zhu et al. found that lower uterine peristaltic wave frequency (<3.0 waves/min) before embryo transfer is associated with higher clinical pregnancy rates in both fresh and frozen-thawed embryo transfer cycles. In a study by Vuong et al. on patients with repeated implantation failure, they found that administering atosiban to patients with uterine peristalsis exceeding 16 waves per 4 minutes could improve pregnancy rates.

Different protocols for endometrial preparation in FET cycles, including natural cycles and hormone replacement therapy (HRT) cycles, create distinct hormonal environments that influence endometrial peristalsis and may impact pregnancy outcomes. Understanding how endometrial peristalsis varies by protocol and its effect on pregnancy outcomes is essential for optimizing IVF strategies.

Therefore, this study aims to evaluate endometrial peristalsis patterns in different FET protocols and their association with pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 - 42 years old
* Scheduled for frozen embryo transfer cycles using hormone replacement therapy protocol or natural cycle protocol (True natural cycles or modified natural cycles)
* Transferred no more than two cleavage embryos or one good-quality blastocyst or no more than two poor-quality blastocysts

Exclusion Criteria:

* Having an allergy and contraindications for exogenous hormone administration (e.g., breast cancer, thromboembolic disease)
* Cycles with preimplantation genetic testing, oocyte donation, or in vitro maturation
* Having untreated uterine or adnexal abnormalities (e.g., intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus, endometrial polyp, large leiomyoma ≥5 cm in diameter, hydrosalpinx, endometrial hyperplasia).
* Use of uterine relaxants or intralipid infusion during the embryo transfer process.
* Use of a GnRH-agonist for downregulation within one month.
* PCOS patients

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women undergoing frozen embryo transfer during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of endometrial peristalsis at different time points, and different FET protocol. | • On the second day to the fourth day of the menstrual cycle in the FET cycles. • The day of progesterone initiation or LH surge/hCG trigger, (before progesterone exposure) • On the day of embryo transfer, immediately prior to the procedure
  Frequency is defined as the number of peristaltic waves per minute.

SECONDARY OUTCOMES:
Direction of peristalsis. | • On the second day to the fourth day of the menstrual cycle in the FET cycles. • The day of progesterone initiation or LH surge/hCG trigger, (before progesterone exposure) • On the day of embryo transfer, immediately prior to the procedure
  Direction of peristalsis is categorized as cervix-to-fundus, fundus-to-cervix, indeterminate, or absent (no contractions observed)
The association between endometrial peristalsis at different time points and pregnancy rates | Up to delivery
  The association between endometrial peristalsis at different time points and pregnancy rates
The correlation between endometrial peristalsis at different time points | • On the second day to the fourth day of the menstrual cycle in the FET cycles. • The day of progesterone initiation or LH surge/hCG trigger, (before progesterone exposure) • On the day of embryo transfer, immediately prior to the procedure
  The correlation between endometrial peristalsis at different time points.
Live birth rates after the one embryo transfer. | At delivery
  Live birth was defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. Live births refer to the individual newborn; for example, a twin delivery represents two live births.
Positive pregnancy test | 10-14 days after embryo transfer
  Defined as serum human chorionic gonadotropin level ≥ 25 mIU/mL.
Clinical pregnancy | 4-6 weeks after embryo transfer
  A pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy.
Ongoing pregnancy | 12 weeks of gestation or beyond
  A pregnancy diagnosed by ultrasonographic or clinical documentation of at least one fetus with a discernible heartbeat at 12 weeks gestation or beyond.
Implantation rate | At 4-6 weeks after embryo transfer
  The number of gestational sacs observed divided by the number of embryos transferred (usually expressed as a percentage).
Ectopic pregnancy | Up to 12 weeks after embryo transfer
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Miscarriage | Up to 22 weeks of gestation
  Spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age, in which the embryo(s) or fetus(es) is/are nonviable and is/are not spontaneously absorbed or expelled from the uterus.
Multiple gestations | At delivery
  A pregnancy with more than one embryo or fetus.
Multiple birth | At delivery
  The complete expulsion or extraction from a woman of more than one fetus, after 22 completed weeks of gestational age, irrespective of whether it is a live birth or stillbirth. Births refer to the individual newborn; for example, a twin delivery represents two births.
Mode of delivery | At delivery
  Vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor).
Birth weight | At delivery
  Weight of the newborn measured right after delivery.
Gestational age at birth | At delivery
  Calculated by gestational age of all live births.
Preterm birth | At delivery
  Defined as delivery at <28, <32, <37 completed weeks. A birth that takes place after 22 weeks and before 37 completed weeks of gestational age.
Gestational diabetes mellitus | At 24-28 weeks of gestation
  A 75-g OGTT, with plasma glucose measurement when the patient is fasting and at 1 and 2 h, at 24-28 weeks of gestation in women not previously diagnosed with diabetes.
Hypertensive disorders of pregnancy | Up to delivery
  Hypertensive disorders of pregnancy: Pregnancy-induced hypertension, pre-eclampsia (early and late), eclampsia, and HELLP syndrome are defined in the American College of Obstetricians and Gynecologists (ACOG) 2020 g
Stillbirth | Up to delivery
  The death of a fetus before the complete expulsion or extraction from its mother after 28 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles. Note: It includes deaths occurring during labor.
Very low birth weight | Up to delivery
  Birth weight less than 1.500 g.
Low birth weight | Up to delivery
  Birth weight less than 2.500 g.
High birth weight | Up to delivery
  Implies growth beyond an absolute birth weight, historically 4.000 g or 4.500 g, regardless of the gestational age.
Very high birth weight | Up to delivery
  Birth weight over 4.500 g for women with diabetes, and a threshold of 5000 g for women without diabetes.
Major congenital abnormalities | Up to delivery
  Structural, functional, and genetic anomalies that occur during pregnancy, and are identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or life-threatening, or cause death. Any congenital anomaly will be included as follows definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
NICU admission | Up to delivery
  The admission of the newborn to the NICU.
Neonatal mortality | Up to delivery
  Death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between 8 and 28 days after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — IVFMD and HOPE Research Center, My Duc Hospital
Locations (2):
- Vietnam (2):
  - My Duc Phu Nhuan Hospital, Ho Chi Minh City
  - IVFMD Phu Nhuan - My Duc Phu Nhuan Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No